CLINICAL TRIAL: NCT01633918
Title: Integrating Internet-supported FeetEnergy Approach in Health Education Lessons to Increase Physical Activity and Reduce Screen Time in Adolescents
Brief Title: FeetEnergy Approach to Increase Physical Activity and Reduce Screen Time in Adolescents
Acronym: FeetEnergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UKK Institute (Other)
Collaborators: Ministry of Education and Culture, Finland (Other)
Responsible Party: Principal Investigator, Minna Aittasalo, Doctor of Health Sciences, UKK Institute
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 166,02
Record Dates: First submitted 2012-06-27; First posted 2012-07-04 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2014-08

CONDITIONS: Physical Activity; Sedentary Behavior; Active Commuting; Psychosocial Factors; Parental Interference
Keywords: intervention; health education; physical activity; sedentary behavior; health promotion; evaluation; RE-AIM
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-supported FeetEnergy approach (Experimental): Schools which integrate Internet-supported approach with two home works in three health education lessons on physical activity
  Interventions: Behavioral: Internet-supported FeetEnergy approach
- Usual health education (Active Comparator): Schools which follow their usual practices in carrying out health education classes on physical activity
  Interventions: Behavioral: Usual health education

INTERVENTIONS:
Behavioral: Internet-supported FeetEnergy approach — Three health education lessons and two homework's about increasing physical activity and reducing screen time
  Arms: Internet-supported FeetEnergy approach
Behavioral: Usual health education — Usual health education lessons
  Arms: Usual health education

SUMMARY:
The purpose of this study is to find out whether an Internet-supported FeetEnergy approach and two home works integrated in three health education lessons can increase adolescents' active commuting to school and leisure-time physical activity and decrease their screen time.

ELIGIBILITY:
Inclusion Criteria:

* student's informed consent and an approval from his/her parent

Exclusion Criteria:

* no informed consent from the student and no approval from his/her parent

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1291 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
change from baseline in meeting physical activity recommendation at 1 month | baseline and 1 month
change from baseline in physical activity recommendation at 7 months | baseline and 7 months
change from baseline in meeting screen time recommendation at 1 month | baseline and 1 month
change from baseline in meeting screen time recommendation at 7 month | baseline and 7 month

SECONDARY OUTCOMES:
change from baseline in psychosocial factors related to physical activity at 1 month | baseline and 1 month
change from baseline in parental interference with physical activity of their child at 1 month | baseline and 1 month
change from baseline in psychosocial factors related to screen time at 1 month | baseline and 1 month
change from baseline in parental interference with screen time of their child at 1 month | baseline and 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Minna M Aittasalo, Dsc, Principal Investigator — UKK Institute
Locations (2):
- Finland (2):
  - Aalto University, Espoo, Aalto
  - The UKK Institute for health Promotion Research, Tampere

REFERENCES:
- [Derived] Aittasalo M, Jussila AM, Tokola K, Sievanen H, Vaha-Ypya H, Vasankari T. Kids Out; evaluation of a brief multimodal cluster randomized intervention integrated in health education lessons to increase physical activity and reduce sedentary behavior among eighth graders. BMC Public Health. 2019 Apr 17;19(1):415. doi: 10.1186/s12889-019-6737-x. PMID 30995905
- [Derived] Jussila AM, Vasankari T, Paronen O, Sievanen H, Tokola K, Vaha-Ypya H, Broberg A, Aittasalo M. KIDS OUT! Protocol of a brief school-based intervention to promote physical activity and to reduce screen time in a sub-cohort of Finnish eighth graders. BMC Public Health. 2015 Jul 10;15:634. doi: 10.1186/s12889-015-2007-8. PMID 26160058
- See also: Related Info — http://www.ukkinstituutti.fi